CLINICAL TRIAL: NCT06965933
Title: Perioperative Use of Erector Spinae Plane Block (ESPB) and Intravenous Lidocaine Infusion in Anesthetic Management of Spinal Surgery in Children
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Maxim Monastirniy, Anesthesiologist-Intensivist, Research Physician, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SaintPetersburgSU
Record Dates: First submitted 2025-04-04; First posted 2025-05-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Regional Anesthesia; Lidocaine Infusion
Keywords: ESPB; Erector Spinae Plane Block; Lidocaine; Regional Anesthesia; Lidocaine infusion; Spinal Surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blockade of the plane straightening the spine (Erector Spinae Plane Block, ESPB). (Experimental)
  Interventions: Procedure: ESP block group
- IV Lidocaine (Active Comparator)
  Interventions: Drug: IV Lidocaine

INTERVENTIONS:
Procedure: ESP block group — The patient will undergo an ESP blockade under the control of ultrasound during the implementation of anesthetic support. A local anesthetic will be injected into the fascial space of the muscles straightening the spine: ropivacaine 0.375%, 3 mg / kg, on both sides.
  Arms: Blockade of the plane straightening the spine (Erector Spinae Plane Block, ESPB).
Drug: IV Lidocaine — During the implementation of anesthetic support, the patient will receive a constant intravenous infusion of lidocaine: a loading dose of 1.5 mg/kg/ h (1 hour), followed by an infusion of 1 mg/kg/h for 24 hours during the perioperative period.
  Arms: IV Lidocaine

SUMMARY:
Testing the hypothesis that in children undergoing spinal surgery, ESP-block will increase the time to emergency anesthesia in the postoperative period compared with intravenous lidocaine infusion.

DETAILED DESCRIPTION:
Interventions for congenital or acquired spinal anomalies are usually voluminous and traumatic, which causes a high level of pain stimulation during the perioperative period. Thus, the problem of pain in spinal surgery is extremely important and is one of the main components of successful treatment.

Combined anesthesia using regional techniques (local anesthesia is added to general anesthesia) can be a significant alternative to performing traditional combined anesthesia with high doses of opioids (narcotic painkillers with undesirable side effects). It allows you to follow the principles of multimodal analgesia, with the possibility of rapid recovery of the patient in the postoperative period.

The use of ESPB (spinal straightening plane blockade) in vertebrology has currently been studied only in adult patients. ESPB is effective and safe for postoperative pain relief after lumbar spine surgery. ESPB can reduce the consumption of opioids (narcotic painkillers) after surgery, increase patient satisfaction, and shorten the length of hospitalization.

Currently, the use of the local anesthetic lidocaine as a medicinal agent for intravenous infusion in children, as an alternative to narcotic anesthesia, is also being actively discussed.

A large number of studies indicate the effectiveness of intravenous lidocaine infusion for perioperative anesthesia in adult patients. In pediatric practice, this technique is not widely used due to the lack of evidence base for efficacy and safety.

Intravenous infusion of lidocaine consistently improves analgesic parameters in the adult and pediatric populations in the first 24 hours, while an effective decrease in the consumption of narcotic painkillers is noted by 48 hours.

Intravenous lidocaine has demonstrated antineuropathic, antihyperalgesic and anti-inflammatory effects and is a new method. Numerous studies in adults have demonstrated the beneficial effects of intravenous lidocaine, including improved pain relief with reduced postoperative use of narcotic painkillers, earlier activation, and shorter length of stay in the intensive care unit. To date, the dose ranges studied in the pediatric population have not been associated with serious side effects, and current evidence suggests that intravenous lidocaine administration will be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Elective surgery on the thoracic and lumbosacral spine. 2. Signed informed consent to participate in the study; 3. Age 3-17 years.

Exclusion Criteria:

1. Contraindications to the use of local anesthetics;
2. Operations on the cervical spine;
3. Contraindications to performing ESPB;
4. The patient's refusal to participate in the study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time before emergency pain relief (opioid). | 24 hours postoperatively
  Time before emergency pain relief (opioid).

SECONDARY OUTCOMES:
the need for opioids in the postoperative period within 24 hours | 24 hours
  the need for opioids in the postoperative period within 24 hours (of the start of anesthesia)
pain level assessment using pain scales (Wong-Baker Faces Pain Rating Scale) | 24 hours postoperatively
  use Wong-Baker Faces Pain Rating Scale (postoperative period)
  The Wong-Baker Faces Pain Rating Scale is used for general assessment of pain intensity in adult patients and children over 3 years of age.
  The scale consists of 6 faces, ranging from laughing (no pain) to crying (unbearable pain).
  Each face corresponds to a certain number of points:
  0 points - a happy smiling face, means no pain (No Hurt); 2 points - a slight smile on the face, means slight soreness (Hurts Little Bit); 4 points - neutral facial expression, means slight pain (Hurts Little More); 6 points - facial expression with slightly furrowed eyebrows, means average pain (Hurts Even More); 8 points - a facial expression with heavily furrowed eyebrows means severe pain (Hurts a Whole Lot); 10 points - a crying, unhappy expression means excessive unbearable pain (Hurts Worst).
assessment of intraoperative analgesia quality (pulse) | during surgery
  pulse monitoring during surgery
assessment of intraoperative analgesia quality (BP) | during surgery
  Blood pressure monitoring during surgery
Complications associated with intravenous lidocaine infusion (general toxic effects on the cardiovascular and central nervous systems) | 24 hours
Complications associated with spinal straightening plane block (ESPB) | 24 hours
  Complications: neurological, bleeding, hematoma, infection.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Sergeevich Monastirniy, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- SaintPetersburgSU, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
By an inappropriate request